CLINICAL TRIAL: NCT00858442
Title: PRP on Children With Retractable Burn Sequelae Who Have Submitted Release of Burn Contractures and Skin Graft on Their Limbs. A Double-Blind Randomized Clinical Trial
Brief Title: Platelet-Rich Plasma (PRP) in Reconstructive Surgery on Children With Retractable Burn Sequelae on Extremities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporation for the Aid of Burned Children (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, maría beatriz quezada, md, Corporation for the Aid of Burned Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-Quezada
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-01

CONDITIONS: Burns
Keywords: Burn sequelae; PRP; Children
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- With PRP (Experimental): Each patient received a single dose of 5cc PRP before the graft.
  Interventions: Procedure: With PRP
- Without PRP (No Intervention): Control patients did not receive any intervention before the graft.

INTERVENTIONS:
Procedure: With PRP — Release of burn contractures and skin graft on the affected limb, a rigorous haemostasis. The surgeon must distribute the activated PRP evenly, forming a very fine clot over it. Immediately the split skin graft must be applied, duly fenestrated. The grafted zone will be measured in it's longest width and length, taking a standardized photograph. On the 5th day the nurse will evaluate the graft's conditions. The evaluation will be done following a previously established follow-up protocol. Measurements of width & length of graft and standardized photo taken at the initiation of the compressive system. Measurement of graft's width & length and standardized photo at the end of the compressive system according protocol. Statistical analysis.
  Arms: With PRP

SUMMARY:
Does the addition of Platelet-Rich Plasma (PRP) to release of burn contractures and skin graft on the limbs of children with retractable burn sequelae reduce the initial time of the compressive treatment and maintain or lower the graft's retraction?

DETAILED DESCRIPTION:
Hypothesis:

1. The use of PRP will allow to initiate sooner the compressive treatment during the post graft surgery evolution, in fewer days on average than the traditional method (18 ds).
2. The use of PRP will maintain the same initial size of the graft. The study's domain corresponds to burn sequelae on children in treatment with reconstructive surgery due to retractile sequelae located on their upper and lower limbs, with functional compromise during their growth process.

One of the treatments used for this problem is the surgical technique of with release of burn contractures and skin graft.

Split skin grafts are at risk of suboptimal "take" due to bleeding and infection which would, on the one hand, delay the initiation of the rehabilitation with preventive compression to avoid the retraction of the grafted area.

20% of the children that arrive in COANIQUEM (approximately 7,000 annually), require rehabilitation. Of these, 32% have surgery and 9% of those are release of burn contractures and skin graft mainly on extremities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with burn sequelae on their upper or lower limbs
* Treated with release of burn contractures and skin graft on their upper or lower limbs
* Between 5 and 21 years old
* Following instructions in their homes
* With informed and written consent
* Weight 35 Kg or more
* Blood count
* Hepatic and coagulation tests
* Paediatric evaluation prior to surgery

Exclusion Criteria:

* Background of blood alterations
* Another current pathology

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2009-03; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M B Quezada, MD, Principal Investigator — Corporation for the Aid of Burned Children
Locations (1):
- Coaniquem, Santiago, Pudahuel, Chile

REFERENCES:
- [Result] Martinez-Zapata MJ, Marti-Carvajal A, Sola I, Bolibar I, Angel Exposito J, Rodriguez L, Garcia J. Efficacy and safety of the use of autologous plasma rich in platelets for tissue regeneration: a systematic review. Transfusion. 2009 Jan;49(1):44-56. doi: 10.1111/j.1537-2995.2008.01945.x. Epub 2008 Oct 14. PMID 18954394
- [Result] Rutkowski JL, Thomas JM, Bering CL, Speicher JL, Radio NM, Smith DM, Johnson DA. Analysis of a rapid, simple, and inexpensive technique used to obtain platelet-rich plasma for use in clinical practice. J Oral Implantol. 2008;34(1):25-33. doi: 10.1563/1548-1336(2008)34[25:AAOARS]2.0.CO;2. PMID 18390240
- [Result] Pietramaggiori G, Scherer SS, Mathews JC, Alperovich M, Yang HJ, Neuwalder J, Czeczuga JM, Chan RK, Wagner CT, Orgill DP. Healing modulation induced by freeze-dried platelet-rich plasma and micronized allogenic dermis in a diabetic wound model. Wound Repair Regen. 2008 Mar-Apr;16(2):218-25. doi: 10.1111/j.1524-475X.2008.00362.x. PMID 18318807
- [Result] Rozman P, Bolta Z. Use of platelet growth factors in treating wounds and soft-tissue injuries. Acta Dermatovenerol Alp Pannonica Adriat. 2007 Dec;16(4):156-65. PMID 18204746
- [Result] Crovetti G, Martinelli G, Issi M, Barone M, Guizzardi M, Campanati B, Moroni M, Carabelli A. Platelet gel for healing cutaneous chronic wounds. Transfus Apher Sci. 2004 Apr;30(2):145-51. doi: 10.1016/j.transci.2004.01.004. PMID 15062754
- [Result] Kazakos K, Lyras DN, Verettas D, Tilkeridis K, Tryfonidis M. The use of autologous PRP gel as an aid in the management of acute trauma wounds. Injury. 2009 Aug;40(8):801-5. doi: 10.1016/j.injury.2008.05.002. Epub 2008 Aug 13. PMID 18703188
- See also: burns scars — http://www.nlm.nih.gov/medlineplus/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited on the day of the scheduled surgery. The researcher checked the inclusion criteria. Explained to the parents and patient surgical procedure, risk of complications and are invited to participate voluntarily in the study. Informed consent is signed. They recruited 44 children in total between April 6,2009 and August 9,2011
Pre-assignment Details: Potential candidates to enter the study were 80. Of these, 20 were excluded for having a weight less than 35 kg; 15 for failing to ensure their attendance at the controls and 1 have coagulation disorders
Groups:
- Without PRP: This arm did not receive any intervention
- With PRP: 4 cc of PRP is evenly distributed before the dermo-epidermic draft.
Period: From Surgery to Start Compression;
Arm/Group | Without PRP | With PRP
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0
Period: Compression:Start to Finish
Arm/Group | Without PRP | With PRP
Started | 21 | 23
Completed | 20 | 20
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: Some patients received more than one graft, as it is shown in result section.
Groups:
- Without PRP: Patients with burns sequelae on their limbs treated with release of burns contractures and skin graft between 2008-2010.
- With PRP: Patients with burns sequelae on their limbs treated with release of burn contractures and skin graft with PRP between 2008-2010.
- Total: Total of all reporting groups
Arm/Group | Without PRP | With PRP | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (3.1) | 14.1 (3.5) | 14.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 13 | 6 | 19
Region of Enrollment [Number; unit: participants]
  Chile | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Median Time Between Surgery Date and Start Date Compression.
Description: Participants were followed from the date of surgery and the date of onset of compression for a minimum of 13.5 days and a maximum of 27 days
Time Frame: day
Population: A participant may have one, two or three areas grafted
Measure: Median (Full Range); unit: day
Units Other Than Participants: grafted area
Groups:
- Without PRP: Patients did not received plasma enrich platelets
- With PRP: Patients received plasma enriched platelets
Arm/Group | Without PRP | With PRP
Number analyzed (Participants) | 19 | 22
Number analyzed (grafted area) | 26 | 33
day | 17 [14 to 24] | 19 [13.5 to 27]
Statistical Analysis 1: Comparison: Without PRP vs With PRP; Test type: Non-Inferiority or Equivalence — Applies normality test of shapiro Wilks = 0.953, P> 0.449 in group without PRP and in PRP group shapiro Wilks=0.946, P > 0.259. The data were normally distributed, with equal variances (Test of levene: F = 0.1234, P> 0.99); p > 0.1574, t-test, 1 sided — Applies t-test for equality of means. t = -1.016 is obtained. p> 0.1574; Mean Difference (Final Values) = -2.452, 95% CI 2-sided [-7.332 to 2.428], Standard Error of Mean 2.452

2. Secondary Outcome: Width of the Graft
Description: Central width measurement graft between the start and the end of the compression
Time Frame: start and end compression
Measure: Median (Inter-Quartile Range); unit: centimeter
Units Other Than Participants: grafted areas
Groups:
- Without PRP: Patients did not receive plasma enriched platelets
Arm/Group | Without PRP | With PRP
Number analyzed (Participants) | 20 | 20
Number analyzed (grafted areas) | 26 | 33
centimeter | 0.1 [-0.25 to 1.35] | 0.3 [-0.5 to 2.05]
Statistical Analysis 1: Comparison: Without PRP vs With PRP; Test type: Non-Inferiority or Equivalence — Applies normality test of shapiro Wilks =0.972, P> 0.687 in group without PRP and in PRP group shapiro Wilks = 0.964, P > 0.410. The data were normally distributed, with equal variances (Test of levene: F = 3.153, P> 0.082); p > 0.593, t-test, 2 sided — Applies t-test for equality of means. t = -0.538 is obtained. p> 0.593; Mean Difference (Final Values) = -0.27186, 95% CI 2-sided [-1.28561 to 0.74189], Standard Error of Mean 0.50519

3. Secondary Outcome: Length of the Graft
Description: Central length measurement graft between the start and the end of the compression
Time Frame: start and end compression
Measure: Median (Inter-Quartile Range); unit: centimeter
Units Other Than Participants: grafted areas
Arm/Group | Without PRP | With PRP
Number analyzed (Participants) | 20 | 20
Number analyzed (grafted areas) | 26 | 33
centimeter | 0.2 [-0.95 to 1.55] | 0.2 [-0.65 to 1.00]
Statistical Analysis 1: Comparison: Without PRP vs With PRP; Test type: Non-Inferiority or Equivalence — Applies normality test of shapiro Wilks=0.822, P<0.001 in group without PRP, and in PRP group shapiro Wilks =0.910, P<0.017. The data were no normally distributed, with equal variances (Test of levene, F=1.324, P>0.255); p > 0.398, Wilcoxon (Mann-Whitney); Mean rank group without PRP= 28.88 Mean rank group with PRP= 26.31 Z value = -0.027

ADVERSE EVENTS:
Time Frame: 2 months
Description: adverse effect is considered the need regrafting bloody small areas.
Arm/Group | Without PRP | With PRP
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Without PRP (N=21) | With PRP (N=23)
regrafting (Surgical and medical procedures) | 1 (1) | 1 (1) — adverse effect is considered the need regrafting bloody small areas

LIMITATIONS AND CAVEATS:
Loss cases: PRP group: 3/23 and group without PRP: 1/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No